CLINICAL TRIAL: NCT02393339
Title: Pre-operative Analgesics for Postoperative Pain Relief After Dental Treatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Avia Fux, pediatric dentist, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0638-14-HMO-CTIL
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Pain, Postoperative; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Study group will receive syrup paracetamol (15 mg/kg) 15 min before the dental treatment
  Interventions: Drug: paracetamol
- controll group (Placebo Comparator): Control group will receive placebo syrup, designed to mimic paracetamol syrup, similar in color and viscosity, 15 min before dental treatment.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: paracetamol — Pre-operative administration of Paracetamol syrup
  Other Names: acetaminophen
  Arms: study group
Drug: placebo — Pre-operative administration of placebo syrup
  Arms: controll group

SUMMARY:
The aim of the study is to compare the efficacy of the pre-operative administration of Paracetamol and placebo in reducing postoperative pain after routine dental treatment in children. This study will be a prospective, placebo-controlled, randomized, double-blind trial. Patients in need of dental treatment with local anesthesia will take part in the study.

Study group will receive syrup paracetamol 15 min before the dental treatment. Control group will receive placebo syrup, similar in color and viscosity, 15 min before dental treatment. the patient, the treating dentist, and the interviewer will be blind to the medication.

Main outcome measure: one of the main investigators will interview the patient at three time points: immediately at the end of the treatment, one hour after taking the pre-operative analgesic and by phone 2.5 hours after taking the pre-operative analgesic. The patient and his parents will be asked if the child is crying (yes/no), complaining about pain (yes/no), needed a different kind of analgesics after the treatment (yes/no). In addition, each child will describe his ⁄ her feelings regarding postoperative pain, using the Wong-Baker Facial Rating Pain Scale

DETAILED DESCRIPTION:
This study will be a prospective, placebo-controlled, randomized, double-blind trial. Patients 5-12 years old, healthy, in need of dental treatment with local anesthesia of Lidocaine 2% with adrenalin 1:100,000 in the Hadassah School of Dental Medicine will take part in the study. The dental treatment will include one of the following procedures: restoration, pulpotomy, pulpectomy, stainless steel crown, extraction. Exclusion criteria: preoperative pain, patients taking analgesics within 5 h prior to the dental treatment, allergic reaction or adverse effect to paracetamol, not available (by phone) at least 2 hours after treatment, patient refuse to drink the syrup.

Study group will receive syrup paracetamol 15 min before the dental treatment. Control group will receive placebo syrup, similar in color and viscosity, 15 min before dental treatment. the patient, the treating dentist, and the interviewer will be blind to the medication.

Data collection: age, gender, type of treatment, type of LA (infiltration /block), time of taking the preoperative analgesic, type of preoperative analgesics ( 1 or 2), time at the end of the treatment and baseline apprehension. Baseline anxiety will be recorded prior to the procedure using Facial Image Scale.

Main outcome measure: one of the main investigators will interview the patient at three time points: immediately at the end of the treatment, one hour after taking the pre-operative analgesic and by phone 2.5 hours after taking the pre-operative analgesic. The patient and his parents will be asked if the child is crying (yes/no), complaining about pain (yes/no), needed a different kind of analgesics after the treatment (yes/no). In addition, each child will describe his ⁄ her feelings regarding postoperative pain, using the Wong-Baker Facial Rating Pain Scale The first two parts of the questionnaire (time 0, 1 h) will be answered in the clinic and the last part (time 2.5 h) by phone; the children will have the scale with the faces with them.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* in need of dental treatment with local anesthesia

Exclusion Criteria:

* preoperative pain,
* patients taking analgesics within 5 h prior to the dental treatment
* allergic reaction or adverse effect to paracetamol
* not available (by phone) at least 2 hours after treatment
* patient refuse to drink the syrup
* dental treatment without local anesthesia

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group | Controll Group
Started | 58 | 56
Completed | 51 | 51
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Controll Group | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.98 (1.53) | 7.08 (1.89) | 7 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 31 | 27 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain, as Measured by Wong-Baker Facial Rating Pain Scale ,After Routine Dental Treatment
Description: This scale measures the unpleasantness or effective dimension of a child's pain experience. The child is shown a set of six cartoon faces with varying facial expressions from smile\laughter to tears. Each face has a numerical value, from 0 (smiling face) to 5 (tears). The child selects the facial expression that best represents his \her experience of discomfort.
Time Frame: 2.5 hours after taking the pre-operative analgesic.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Controll Group
Number analyzed (Participants) | 51 | 51
Participants
  Wang-Baker Scale 0 | 20 | 20
  Wang-Baker Scale 1 | 7 | 11
  Wang-Baker Scale 2 | 10 | 9
  Wang-Baker Scale 3 | 5 | 3
  Wang-Baker Scale 4 | 0 | 2
  Wang-Baker Scale 5 | 9 | 6

ADVERSE EVENTS:
Time Frame: 3.5 hours
Arm/Group | Study Group | Controll Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02393339/Prot_SAP_000.pdf